CLINICAL TRIAL: NCT05968157
Title: MIRAI-MRI: Comparing Screening MRI for Patients at High Risk for Breast Cancer Identified by Mirai and Tyrer-Cuzick
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Massachusetts Institute of Technology (Other); Breast Cancer Research Foundation (Other)
Responsible Party: Principal Investigator, Mohammad Salman Shazeeb, Director - Image Processing & Analysis Core; Director of Preclinical MRI & Co-Director of Scientific Affairs (Advanced MRI Center); UMass Chan Medical School, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY000000485; MIT_s5822 (Other Grant/Funding Number: Massachusetts Institute of Technology Subaward); SPEC-22-015 (Other Grant/Funding Number: Breast Cancer Research Foundation)
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Screening; Artificial Intelligence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- High Risk Participants--MIRAI (Experimental): Patients who are deemed high risk on standard breast screening mammogram by the MIRAI model
  Interventions: Diagnostic Test: Breast MRI; Device: MIRAI
- High Risk Participants--non-MIRAI (Active Comparator): Patients who are deemed high risk by Tyrer-Cuzick model but not MIRAI
  Interventions: Diagnostic Test: Breast MRI

INTERVENTIONS:
Diagnostic Test: Breast MRI — Supplemental MRI (in addition to standard of care MRI).
Device: MIRAI — Artificial intelligence software
  Arms: High Risk Participants--MIRAI

SUMMARY:
Accurate risk assessment is essential for the success of population screening programs and early detection efforts in breast cancer. Mirai is a new deep learning model based on full resolution mammograms.

Mirai is a mammography-based deep learning model designed to predict risk at multiple timepoints, leverage potentially missing risk factor information, and produce predictions that are consistent across mammography machines. Mirai was trained on a large dataset from Massachusetts General Hospital (MGH) in the United States and found to be significantly more accurate than the Tyrer-Cuzick model, a current clinical standard.

The primary aim of this study is to prospectively quantify the clinical benefit (i.e. MRI/CEM cancer detection rate) of Mirai-based guidelines and to compare them to the current standard of care.

1. Conduct a prospective study where patients who are identified as high risk by Mirai guidelines are invited to receive supplemental MRI within 12 months.
2. Compare cancer outcomes between patients only identified as high risk by Mirai and patients identified as high risk by existing guidelines The secondary aim is to study the impact of new guidelines by race and ethnicity, to ensure equitable improvements in cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Women who were identified as high risk on the retrospective study (dating from 2017-2025) using MIRAI will be recruited and consented for the prospective study
* Women over 40 years of age identified as high risk according to traditional guidelines will also be potentially eligible for this study
* Following consent and enrollment in the study, a participant will subsequently receive the following:

  1. These patients will be invited to receive a supplemental MRI examination currently considered the most sensitive test for breast cancer detection.
  2. Any positive diagnosis on MRI will be followed by biopsy to confirm 'truth" of diagnosis.
* To be selected, a given record must include the following:

  1. A report of a routine screening mammogram or diagnostic mammogram, and availability of the DICOM images from that report with the PACS system.
  2. Reports of all follow up screening and diagnostic studies documented on PACS.
  3. Some may have interventional procedures (as long as all of these are done at one of Umass sites) and documentation of these biopsy results in the hospitals EHR.

Exclusion Criteria:

* Under age 40. Women under 40 years are not routinely xrayed with a mammogram.
* Xray breast cancer screening imaging study that has artifacts, corruption, or other image quality degradation.
* Pregnant patients because they do not routinely receive screening mammogram
* Adult male patients with breast cancer

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-04 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
CDR Mirai Assessment versus CDR Traditional High Risk Screening | 1.5 years (duration of patient recruitment and outcome data collection)
  Cancer detection rate from breast MRI following Mirai assessment of high risk on a screening mammogram performed less than 1 year ago and compared with established CDR in traditional high risk screening.

SECONDARY OUTCOMES:
Cancer development within study population versus general population of average risk women | 1.5 years (duration of patient recruitment and outcome data collection)
  On subsequent follow-up with standard of care, assessment of what percentage of the study population develops breast cancer as compared to the general population of women at average risk of breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Salman Shazeeb, PhD, Principal Investigator — UMass Chan Medical School
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No